CLINICAL TRIAL: NCT05435703
Title: The Effect of Renal Cysts on Laboratory Diagnostics of Primary Aldosteronism
Brief Title: Renal Cysts and Primary Aldosteronism
Status: Completed | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); Kuopio University Hospital (Other); Tampere University (Other)
Responsible Party: Sponsor
Other Study IDs: R20023
Record Dates: First submitted 2021-04-30; First posted 2022-06-28 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Primary Aldosteronism
Keywords: Adrenal vein sampling; Renal cysts; Renin concentration; Renin activity
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During routine subtyping of confirmed primary aldosteronism by adrenal vein sampling extra plasma samples are drawn from both renal veins and from inferior vena cava. Plasma renin concentration and renin activity are analysed from these samples. Adrenal computed tomographies are analysed for cysts and other possible pathology by a blinded radiologist. Aim is to evaluate correlation between renal pathology and renin measurements.

DETAILED DESCRIPTION:
Aim of the study is to evaluate the prevalence of renal cysts and their association with renin concentrationand acitivity in samples from renal veins and inferior vena cava (IVC) in patients who undergo an adrenal vein sampling (AVS) because of primary aldosteronism.

In a prospective study up to 200 patients who have been referred to Tampere University Hospital for AVS are recruited during 24 months. Informed consent is taken. Clinical, medication, radiological and laboratory information according to Endcrine Society guidelines is collected. Interventional radiologist will draw venous blood from both renal veins and from IVC for later renin analyses. One, blinded radiologist will record renal pathology of cysts but also other abnormal radiologic features.

An interim analysis will be done when 60-100 patients have been recruited or at 6-12 months from the start of the study. Study will be stopped if significant difference can be found in renin measurement in patients with renal cysts compared with patients without renal cysts.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed primary aldosteronism according to Endocrine Society guidelines
* Adrenal vein sampling performed in Tampere University Hospital
* Informed consent

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with confirmed primary aldosteronism undergoing subtyping by adrenal vein sampling
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Association of any renal cyst finding to graded baseline renin concentration (mU/L) | Baseline
  Number of patients with renal cysts when renin concentration (mU/L) is low, low normal or high normal to high

SECONDARY OUTCOMES:
Correlation of renin concentration (mU/L) in inferior vena cava in all patients and in patients with or without renal cysts (or other renal pathology) | During procedure
  Renin concentration difference (mU/L)
Correlation of renin activity (ng of Ang I/ml/h) in inferior vena cava in all patients and in patients with or without renal cysts (or other renal pathology) | During procedure
  Renin activity difference (ng of Ang I/ml/h)
Correlation of renin concentration (mU/l) in right and left renal vein from the side with or without renal cysts (or other renal pathology) | During procedure
  Concentration difference (mU/l)
Correlation of renin activity (ng of Ang I/ml/h) in right and left renal vein from the side with or without renal cysts (or other renal pathology) | During procedure
  Activity difference (ng of Ang I/ml/h)
Prevalence (%) of renal cysts in patients in computed tomography with contrast media | Baseline
  Prevalence of cysts
Association of prevalence of renal cysts (%) with severity of hypertension | Baseline
  Percentage of patients with renal cysts when patients are grouped according to quartiles of severity of hypertension
Association of prevalence of renal cysts (%) with duration (years) of hypertension | Baseline
  Percentage of patients with renal cysts when patients are grouped according to quartiles of duration of hypertension (years)
Association of prevalence of renal cysts (%) with plasma potassium concentration (mmol/l) | Baseline
  Percentage of patients with renal cysts (%) when patients are grouped according to quartiles of lowest plasma potassium
Association of prevalence of renal cysts (%) with severity of primary aldosteronism | Baseline
  Percentage of patients with renal cysts when patients are grouped according to quartiles of aldosterone to renin ratio (pmol/L)/(mU/L)
Renin concentration (mU/l) in renal veins on the side of renal cysts compared with the side with no cysts of each kidney | During procedure
  Concentration difference
Renin concentration (mU/l) in inferior vena cava in patients with renal cysts compared with patients with no cysts | During procedure
  Concentration difference
Renin activity (ng of Ang I/ml/h) in renal veins on the side of renal cysts compared with the side with no cysts | During procedure
  Activity difference
Renin activity (ng of Ang I/ml/h) in inferior vena cava in patients with renal cysts | During procedure
  Activity difference
Association of renal cyst finding to baseline renin concentration (mU/l) in different age groups | Baseline
  Number of patients with renal cysts when renin concentration is low, low normal or high normal to high

CONTACTS AND LOCATIONS:
Overall Officials: Pasi I Nevalainen, MD, PhD, Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: Undecided
IPD may not be shareable according to local laws and regulations